CLINICAL TRIAL: NCT02615496
Title: Evaluation of Physician and Patient Knowledge of Safety and Safe Use Information for Aflibercept in Europe: An Observational Postauthorisation Study
Brief Title: Evaluation of Physician and Patient Knowledge of Safety and Safe Use Information for Aflibercept
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: RTI Health Solutions (Other)
Responsible Party: Sponsor
Other Study IDs: 16526; EY1301 (Other: Company internal)
Record Dates: First submitted 2015-10-21; First posted 2015-11-26 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Macular Degeneration
Keywords: Health Care Surveys; Vascular Endothelial Growth Factor
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Educational materials: Physicians
  Interventions: Behavioral: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321)
- Educational materials: Patients
  Interventions: Behavioral: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321)

INTERVENTIONS:
Behavioral: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321) — Survey to measure physician awareness and understanding of the key messages in the educational materials: the prescriber guide and video.
  Groups: Educational materials: Physicians
Behavioral: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321) — Survey to measure patient awareness and understanding of the key messages in the educational materials: the patient booklet "Your guide to EYLEA," patient information leaflet, and audio CD.
  Groups: Educational materials: Patients

SUMMARY:
The study will be an observational, cross-sectional study of knowledge, understanding, and self-reported behavior among a sample of physicians and patients with recent aflibercept experience in a total of up to five European countries.

ELIGIBILITY:
Inclusion Criteria:

Physicians eligibility:

* Licensed and practicing ophthalmologist
* Prescribed and administered aflibercept to at least one patient in the past 6 months

Patients eligibility:

* Patient has been administered aflibercept at least once within the last 6 months for any indication and is returning for a subsequent visit.
* Patient is aged 18 years or older.
* Patient is able to understand and sign the consent form and patient questionnaire.
* Patient can understand the native language of the country in which the study is being conducted.
* Patient has not participated in a clinical trial for the treatment of an aflibercept indication (e.g., wAMD, CRVO, or DME) in the past 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Physicians eligible to participate will be ophthalmologists who have administered aflibercept in the past 6 months.
  Patients eligible to participate will be those who have already received at least one aflibercept injection and are returning for a subsequent visit. Patients will be aged 18 years or older, and will be able to understand the native language of the country in which the study is conducted.
Sampling Method: Non-Probability Sample
Enrollment: 716 (Actual)
Dates: Start 2015-12-07 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
The proportion of physicians with accurate knowledge and understanding of key safety information (identified risks and prescribing behaviors) contained in the Eylea educational materials as assessed by a study specific questionnaire. | Up to 2 years
The proportion of patients with accurate knowledge and understanding of key safety information (identified risks and guidelines) contained in the Eylea educational materials as assessed by a study specific interviewer administered questionnaire. | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (5):
- Many Locations, France
- Many Locations, Germany
- Many Locations, Italy
- Many Locations, Spain
- Many Locations, United Kingdom